CLINICAL TRIAL: NCT06257069
Title: Tremor Retrainer Software Application for Functional Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Child Neurology Foundation (Unknown)
Responsible Party: Principal Investigator, Jordan F Garris, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230161
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Functional Movement Disorder; Functional Neurological Disorder; Functional Neurological Symptom Disorder
Keywords: Functional Tremor
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): All subjects will receive intervention with Tremor Retrainer smartphone application
  Interventions: Device: Tremor Retrainer Smartphone Application

INTERVENTIONS:
Device: Tremor Retrainer Smartphone Application — The Tremor Retrainer smartphone application uses the smartphone's built-in accelerometer to calculate a patient's tremor frequency when the smartphone is strapped to the patient's wrist. The application will provide auditory cues to the patient with a treatment frequency at 2/3 the patient's baseline tremor frequency for half a session, then 1/3 the patient's baseline tremor frequency for the second half of the session. Meanwhile, oscillatory movements will be continuously analyzed with frequency calculated and displayed relative to goal frequency, so that the patient receives continuous feedback via a visual dial as to whether they are meeting treatment goals. Intervention will consist of a one-week Tremor Retrainment Protocol.

SUMMARY:
The purpose of this clinical trial is to learn about the Tremor Retrainer smartphone application and Simplified Functional Movement Disorder Rating Scale in patients with functional tremor. The main questions the study aims to answer are:

1. Is the Tremor Retrainer application usable for patients and are there signs that it can help functional tremor?
2. Can a televideo administration of the Simplified Functional Movement Disorder Rating Scale give enough information to use this scale via televideo in future studies?

DETAILED DESCRIPTION:
Following a one-week observation period, 20 subjects will complete the one-week four hour Tremor Retrainer smartphone protocol.

The study will consist of 4 in-person visits over 3-4 months and one televideo visit the same day as study visit 1.

For Objective 1, the investigators will evaluate mHealth Application Usability Questionnaire scores after subjects complete Tremor Retrainer protocol and compare Simplified Functional Movement Disorder Rating Scale (S-FMDRS) scores before (study visit 2) and after (study visits 3 and 4) intervention between groups.

For Objective 2, the investigators will evaluate which components can be scored after televideo administration of S-FMDRS and measure correlation between randomly-ordered sequential in-person and televideo S-FMDRS administration.

For Objective 3, the investigators will measure change and variability in S-FMDRS between study visit 1 and 2. S-FMDRS scoring will be completed via video review by a movement disorder neurologist blinded to timing of visit relative to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10 years and older, any gender, any race
2. Functional tremor as defined by Espay and Lang25, diagnosed by a movement disorders neurologist, involving at least 1 arm and ongoing at time of enrollment.
3. Access to internet and a laptop or tablet with a videocamera.
4. Informed consent obtained and signed
5. Subject understands study procedures and is able to comply with study procedures for duration of study

Exclusion Criteria:

1. Parkinson's disease, essential tremor, or other disorders causing involuntary movements in addition to functional tremor
2. Cognitive impairment with previously diagnosed intellectual disability (IQ<70) or dementia
3. Hearing impairment not addressed by hearing aids
4. Prior enrollment in clinical trial involving the Tremor Retrainer application

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
mHealth Application Usability Questionnaire | Study visit 3
  Usability Questionnaire. Score range: 21-147 with higher scores indicating better usability
Simplified Functional Movement Disorder Rating Scale | Study visits 1-4
  Videorecorded severity scale. Score range: 0-54 with higher scores indicating greater severity (worse movements)

OTHER OUTCOMES:
Adherence | Study visit 3
  Duration of sessions completed
Clinical Global Impression Severity Scale - Clinician Rated | Study visits 1-4
  Clinician rated impression of tremor severity. Score range: 1-7, with 7 being most severely affected
Clinical Global Impression Improvement Scale - Clinician Rated | Study visits 2-4
  Clinician rated impression of tremor change. Score range: 1-7, with 1 being best and 7 being worst.
Clinical Global Impression Improvement Scale - Patient Rated | Study visits 2-4
  Patient rated impression of tremor change. Score range: 1-7, with 1 being best and 7 being worst.
Visual Analog Scale | Between study visits 2-3
  Patient rated impression of tremor severity. Score range: 0-10, with 10 being worst tremor imaginable.
36-Item Short-Form Survey | Study visits 1 and 4
  Quality of life scale. Score range: 0-100, with 100 being best.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Garris, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data, including raw scores of outcome measures will be available for review.
Supporting Information: Study Protocol, SAP
Time Frame: Data anticipated to be available in 2026.
Access Criteria: Anonymized participant data will be publicly available.
URL: https://www.ithriv.org/ithriv-research-data-commons